CLINICAL TRIAL: NCT02922179
Title: Descriptive Analysis of Long- and Intermediate-Acting Insulin in Adult Diabetics
Status: Completed | Type: Observational
Sponsor: Biologics & Biosimilars Collective Intelligence Consortium (Other)
Collaborators: HealthCore, Inc. (Industry); Aetna, Inc. (Industry); University of Alabama; Rheumatologist and Healthcare Research (Unknown); AbbVie (Industry); Amgen (Industry); Boehringer Ingelheim (Industry); Kaiser Permanente (Other); Harvard Pilgrim Health Care (Other); Merck Sharp & Dohme LLC (Industry); Momenta Pharmaceuticals, Inc. (Industry); Pfizer (Industry); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: BBCIC Insulins
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Diabetes
Keywords: Insulin; Diabetes; Biologic and Biosimilars Collective Intelligence Consortium; BBCIC; Descriptive analysis
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes Type 1: Individuals diagnosed with type 1 diabetes exposed to Long- and intermediate- acting insulins
  Interventions: Drug: Long- and intermediate- acting insulins
- Diabetes Type 2: Individuals diagnosed with type 2 diabetes exposed to Long- and intermediate- acting insulins
  Interventions: Drug: Long- and intermediate- acting insulins

INTERVENTIONS:
Drug: Long- and intermediate- acting insulins — alone or in combination with metformin, short-acting insulin, or second-generation sulfonylurea
  Other Names: NPH, Lantus, Levemir, Toujeo

SUMMARY:
Over the past 40 years, new types of insulins have been marketed to mirror the effect of endogenous insulin. With the existing long-acting insulin product patents expiring and the FDA approval of new biosimilar and innovator insulins, adults with diabetes and their physicians will have additional therapeutic options. This observational study will describe the patient characteristics of new and existing users of long-acting or intermediate acting insulins with and without oral anti-diabetic agents (OAD) as well as acute hypoglycemic episodes, acute cardiac events, and A1C measures. The Biologic and Biosimilars Collective Intelligence Consortium (BBCIC) will use the findings from this descriptive analysis to design a comparative study evaluating the real-world effectiveness and safety of biosimilar and innovator insulins.

DETAILED DESCRIPTION:
Additional information:

This protocol was designed as a descriptive analysis, not to support a hypothesis. This information is being provided to the public in the interest of transparency and for demonstrating the BBCIC's Distributed Research Network's (DRN) ability to define exposures, outcomes, covariates and confounders. When published, the report will caution that the protocol does not support any ability to compare safety or effectiveness but instead is to be used only to explore the feasibility of future, more detailed comparative analyses and to better understand the capabilities of the BBCIC project. Further, the report will caution that information from this protocol should not affect use of the medical products described in any way and the fact that the BBCIC is performing this descriptive analysis in no way suggests there is a safety or effectiveness issue with any of the products described.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with baseline period of 183 days with continuous medical and pharmacy coverage preceding the first prescription fill
* new and current users of the following exposures

  * Long-acting insulin (insulin detemir, glargine) alone or with metformin (LAI)
  * Long-acting insulin (insulin detemir, glargine) plus rapid/short acting insulin (with or without metformin) (LAI+R)
  * Long-acting insulin (insulin detemir, glargine) plus second-generation sulfonylurea agent (Glimepiride, Glipizide, Glipizide/Metformin, Glyburide, Glyburide/Metformin) (with or without metformin) (LAI+sulfa)
  * NPH insulin (Humulin, Novolin) alone or with metformin (NPH)
  * NPH insulin (Humulin, Novolin) plus rapid/short acting insulin (with or without metformin) (NHP+R)
  * NPH insulin (Humulin, Novolin) plus second-generation sulfonylurea agent (Glimepiride, Glipizide, Glipizide/Metformin, Glyburide, Glyburide/Metformin (with or without metformin) (NPH + sulfa)

Exclusion Criteria:

* Adult patients with diabetes with health insurance evidence of insulin pumps and/ or insulin pump supplies, gestational diabetes, liver disorders, dialysis, end-stage renal disease (ESRD), amputations, hemoglobinopathy, hemolytic anemia, or sickle cell anemia or transfusion
* Emergency Department (ED) visit for hypoglycemia; hospitalization or ED visit for cardiovascular event (stroke, acute myocardial infarction, unstable angina or diagnosis consistent with unstable angina -- i.e., occlusion without infarction or coronary insufficiency).
* Adult patients with diabetes on any other insulins except cohort insulins (i.e., rapid/short unless in combinations above).*
* Adult patients with diabetes on first-generation sulfonylureas, Dipeptidyl peptidase-4 (DPP4), Glucagon-like Peptide (GLP), Sodium-glucose cotransporter-2 (SGLT-2) or Thiazolidinediones (TZD) agents, alone or in combination with cohort defining drugs*:

  * First generation sulfonylurea agents (chlorpropamide, tolazamide )
  * TZDs (pioglitazone, pioglitazone/metformin, rosiglitazone, rosiglitazone/metformin
  * DPP4s (sitagliptin, saxagliptin, linagliptin, alogliptin)
  * GLP1 (exenatide, liraglutide, dulaglutide)
  * SGLT-2 (empagliflozin, canagliflozin, dapagliflozin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects are selected according to inclusion criteria from a source population within the Sentinel Common Data Mode v5.0.1 (SCDM). The SCDM includes over 100 million individuals with 358 million person-years of observation time who are covered by Aetna, Anthem, Group Health Cooperative, Harvard Pilgrim Health Care, and HealthPartners. The time period assessed will be 1/1/2011 - 9/30/2015.
Sampling Method: Non-Probability Sample
Enrollment: 103951 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
serious hypoglycemic events | Anticipated completion January 2017
  Incidence of serious hypoglycemic events in adult patient with diabetes population who use long- or intermediate-acting insulin

SECONDARY OUTCOMES:
Serious cardiac events | Anticipated completion January 2017
  Incidence of serious cardiac events in adult patient with diabetes population who use long- or intermediate-acting insulin

OTHER OUTCOMES:
A1C control | Anticipated completion January 2017
  A1C control in adult patient with diabetes population who use long- or intermediate-acting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Dan Kent, PharmD,CDE, Principal Investigator — Kaiser Permanente; Cheryl Walraven, PhD, Principal Investigator — Aetna, Inc.

IPD SHARING:
Plan to Share IPD: Yes
BBCIC Charter requires transparency and publication
Supporting Information: SAP

REFERENCES:
- [Result] Kent DJ, McMahill-Walraven CN, Panozzo CA, Pawloski PA, Haynes K, Marshall J, Brown J, Eichelberger B, Lockhart CM. Descriptive Analysis of Long- and Intermediate-Acting Insulin and Key Safety Outcomes in Adults with Type 2 Diabetes Mellitus. J Manag Care Spec Pharm. 2019 Nov;25(11):1162-1171. doi: 10.18553/jmcp.2019.19042. Epub 2019 Aug 12. PMID 31405345
- [Result] McMahill-Walraven CN, Kent DJ, Panozzo CA, Pawloski PA, Haynes K, Marshall J, Brown J, Eichelberger B, Lockhart CM. Harnessing the Biologics and Biosimilars Collective Intelligence Consortium to Evaluate Patterns of Care. J Manag Care Spec Pharm. 2019 Nov;25(11):1156-1161. doi: 10.18553/jmcp.2019.19041. Epub 2019 Aug 9. PMID 31397619
- See also: The Biologics and Biosimilars Collective Intelligence Consortium (BBCIC) was established in 2015 to address anticipated needs for post-marketed evidence generation for novel biologics, their corresponding biosimilars and other related products. — http://bbcic.org